CLINICAL TRIAL: NCT04666233
Title: Does Personal Protective Equipment for the Prevention of SARS-Cov-2 Infection Impact the Timing of Ventilation in Neonates Needing Resuscitation at Birth? A Crossover Randomized Controlled Trial
Brief Title: Personal Protective Equipment for the Prevention of SARS-Cov-2 During Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SARS-CoV-2-NEO-Res-01
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Neonates Needing Resuscitation at Birth

STUDY DESIGN:
Masking Description: The statistician performing data analysis will be masked to treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resuscitation with PPE for prevention of SARS-Cov-2 infection (Experimental)
  Interventions: Procedure: Neonatal resuscitation with PPE for the prevention of SARS-Cov-2 infection
- Resuscitation without PPE for prevention of SARS-Cov-2 infection (Active Comparator)
  Interventions: Procedure: Neonatal resuscitation without PPE for the prevention of SARS-Cov-2 infection

INTERVENTIONS:
Procedure: Neonatal resuscitation with PPE for the prevention of SARS-Cov-2 infection — The team will perform neonatal resuscitation with PPE for the prevention of SARS-Cov-2 infection
  Arms: Resuscitation with PPE for prevention of SARS-Cov-2 infection
Procedure: Neonatal resuscitation without PPE for the prevention of SARS-Cov-2 infection — The team will perform neonatal resuscitation without PPE for the prevention of SARS-Cov-2 infection
  Arms: Resuscitation without PPE for prevention of SARS-Cov-2 infection

SUMMARY:
There has been an increasing number of SARS-CoV-2 infections in pregnant women and neonates. Interventions including open airway suctioning, positive pressure ventilation, non-invasive respiratory support, tracheal intubation, and endotracheal drug administration are aerosol-generating medical procedures and may create a risk to the unprotected healthcare providers. The impact of using personal protective equipment during neonatal resuscitation maneuvers is unknown.

The objective of this study will be to compare the beginning of PPV and the duration of intubation between performing resuscitation with PPE for the prevention of SARS-Cov-2 infection and resuscitation without PPE for the prevention of SARS-Cov-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Level III neonatal intensive care unit consultants, pediatric residents, and nurses. Participants will be divided into teams including a consultant and a nurse or a resident and a nurse during the simulation.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Initiation of positive pressure ventilation | 5 minutes

SECONDARY OUTCOMES:
Duration of intubation procedure | 5 minutes
Correct use of personal protective equipment | 20 minutes
Participant's opinion on discomfort using personal protective equipment | 20 minutes
  Level of discomfort in performing the procedures: 0 (no discomfort), 1 (low discomfort) ,2 (high discomfort)
Time of initiation of chest compressions | 20 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Central Teaching Hospital of Bolzano/Bozen, Bolzano
  - Daniele Trevisanuto, Padua

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Watson CM, Duval-Arnould JM, McCrory MC, Froz S, Connors C, Perl TM, Hunt EA. Simulated pediatric resuscitation use for personal protective equipment adherence measurement and training during the 2009 influenza (H1N1) pandemic. Jt Comm J Qual Patient Saf. 2011 Nov;37(11):515-23. doi: 10.1016/s1553-7250(11)37066-3. PMID 22132664
- [Result] Trevisanuto D, Moschino L, Doglioni N, Roehr CC, Gervasi MT, Baraldi E. Neonatal Resuscitation Where the Mother Has a Suspected or Confirmed Novel Coronavirus (SARS-CoV-2) Infection: Suggestion for a Pragmatic Action Plan. Neonatology. 2020;117(2):133-140. doi: 10.1159/000507935. Epub 2020 Apr 24. PMID 32335559
- [Result] Aziz K, Lee HC, Escobedo MB, Hoover AV, Kamath-Rayne BD, Kapadia VS, Magid DJ, Niermeyer S, Schmolzer GM, Szyld E, Weiner GM, Wyckoff MH, Yamada NK, Zaichkin J. Part 5: Neonatal Resuscitation: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S524-S550. doi: 10.1161/CIR.0000000000000902. Epub 2020 Oct 21. No abstract available. PMID 33081528
- [Derived] Cavallin F, Lupi F, Bua B, Bellutti M, Staffler A, Trevisanuto D. Impact of personal protective equipment on neonatal resuscitation procedures: a randomised, cross-over, simulation study. Arch Dis Child Fetal Neonatal Ed. 2022 Mar;107(2):211-215. doi: 10.1136/archdischild-2021-322216. Epub 2021 Sep 6. PMID 34489350